CLINICAL TRIAL: NCT01380470
Title: Prevalence of Undiagnosed Sufferers in Murcia :Cross-sectional Study
Brief Title: Prevalence of Undiagnosed Chronic Obstructive Pulmonary Disease Sufferers in the Region of Murcia
Status: Completed | Type: Observational
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: MurciaSalud (Other Government); Public Health Service, Murcia (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: Brisa I
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Diagnosis differential; Dyspnea/classification; Dyspnea/etiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: Group of patients seen in consultation not previously diagnosed with COPD, both sexes, aged between 40 and 70 years.

SUMMARY:
The purpose of this study is determine the prevalence of undiagnosed Chronic Obstructive Pulmonary Disease (COPD) in population served and with exposure to cigarettes in the Region of Murcia

DETAILED DESCRIPTION:
COPD is a serious, chronic and very disabling, associated with smoking and aging. Therefore it is a preventable and treatable process. It is know to be a pathology under diagnosed and when diagnosis, this is done in advanced stage, resulting to rise to more complication and more severe, in a addition to a high social and economic cost.

Therefore, take out an epidemiological study, observational, multicentre, whose main objective is estimate the prevalence of undiagnosed COPD in population served between 40 and 70 years and exposure to cigarettes in the Region of Murcia.

Other objectives are estimate the proportion of patients already diagnosed, identifying risk factors associated with not previous diagnosis of COPD and describe the history of symptoms in them. Description of therapeutic manage and motivation to give up smoking.

The study was carried out with 120 researcher doctors and 120 researcher nurses from 40 health centers in the Region of Murcia.

Each researcher will select 10 patients for the main objective and 10 for objectives related to manage of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40 and 70 years of both sexes
2. With a history of smoking (current or past)
3. Do not diagnosed with COPD at the time of completion of study

Exclusion Criteria:

1. Prior diagnosis of COPD or Asthma
2. A condition prevents performing spirometry
3. Patients displaced

For those diagnosed with COPD:

Inclusion Criteria:

* Subject treated in CS there is explicit evidence for the disease

Exclusion Criteria:

* Subjects who at the time of the consultation arouse suspicion of previously undiagnosed COPD

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group of patients seen in consultation not previously diagnosed with COPD, both sexes, aged between 40 and 70 years.
Sampling Method: Probability Sample
Enrollment: 1052 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC,Forced Expiratory Volume 1/ Forced Vital Capacity | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Asensio Lopez Santiago, MD, Principal Investigator — Consejeria de sanidad y consumo, Direccion general de planificacion, ordenacion sanitaria y farmaceutica e investigacion.
Locations (1):
- Fundación para la Formación e Investigación Sanitarias de la Región de Murcia, Murcia, Murcia, Spain